CLINICAL TRIAL: NCT04492228
Title: Randomized Open Controlled Clinical Trial to Evaluate the Effectiveness of a Eucaloric Ketogenic Nutrition in Comparison With a Standard Nutrition in Covid-19 Disease in Reducing Cytokine Storm Syndrome and ARDS
Brief Title: Eucaloric Ketogenic Diet in COVID-19 Cytokine Storm Syndrome
Acronym: ketocovidiet
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ospedale Policlinico San Martino (Other)
Responsible Party: Principal Investigator, Sukkar Samir, MD, Dr Samir Giuseppe Sukkar, Ospedale Policlinico San Martino
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KETOCOV-1
Record Dates: First submitted 2020-07-25; First posted 2020-07-30 (Actual); Last update posted 2020-09-30 (Actual); Status verified 2020-09

CONDITIONS: Covid19; Ketogenic Dieting
MeSH Terms: conditions — COVID-19 | interventions — Diet, Ketogenic

STUDY DESIGN:
Intervention Model Description: This is a controlled, randomized, open-label, clinical trial designed to determine whether a ketogenic diet,in comparison with a standard diet, improves mortality and reduces ventilator requirements or ICU access in patients with coronavirus disease.
  The study team will prospectively enroll 50 patients with COVID-19 infection administering a 4:1 ratio ketogenic formula (both enteral or parenteral) and 50 with standard diet
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ketogenic diet group (Experimental): patients with COVID-19 feeding with a ketogenic diet (4.1 formula)
  Interventions: Other: Ketogenic diet
- Standard diet group (No Intervention): patients with COVID-19 feeding with a standard diet

INTERVENTIONS:
Other: Ketogenic diet — Eucaloric Ketogenic diet % composition : protein (27%), lipids (67%), carbohydrates (6%: <30g/day). In pts in artificial nutrition : Eucaloric Ketogenic parenteral nutrition % composition : aminoacids (27%), lipids (67%), carbohydrates (6%: <30g/day)
  Arms: Ketogenic diet group

SUMMARY:
Covid 19 pandemia is causing millions of deaths worldwide. To date, the evidence gathered suggests that the subgroup of patients who present the most serious clinical feature of COVID-19 could have a "cytokine storm syndrome" better defined as secondary hemophagocytic lymphohistiocytosis (sHLH), characterized by acute respiratory distress (ARDS) and septic shock, followed by multi-organ failure due to an excess of cytokines induced by the inflammatory response to the virus.

The reduction of phagocytic hyperactivation represents a possible treatment for HLH.

Lowering the availability of glucose, the only substrate of aerobic glycolysis and of the Warburg effect in activated macrophages, through the use of ketogenic diets could be a promising solution.

Actually diet is not recognized as impacting on the evolution of COVID-19, however, scientific literature data show that a low carbohydrate and high lipid diet (ketogenic diet) can inhibit inflammation and lead to a clinical improvement of respiratory function.

The hypothesis of this study is that the administration of a ketogenic diet could improve mortality, lower the access to ICU and the need of NIV.

The plan is to enroll 50 patients with COVID 19 infection and administer a 1:4 ketogenic formula during hospitalization in order to verify these outcomes.

ELIGIBILITY:
Inclusion Criteria:

* documented clinical diagnosis of COVID-19 supported by clinical features and by the positivity to at least one pharyngeal swab
* age ≥18 years
* informed written consent

Exclusion Criteria:

* Type I diabetes
* Type II diabetes in therapy with insulin, sulphonylureas, repaglinide, GLP-1 analogues, SGLT2 inhibitors
* Recent acute cardiovascular event (within a month)
* Food allergies to diet components
* Any metabolic disorder capable of influencing gluconeogenesis
* Clinical history of severe hypertriglyceridemia with or without pancreatitis
* Pregnancy and/or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2020-09-01 (Actual); Primary Completion 2020-12-31 (Estimated); Study Completion 2021-05-30 (Estimated)

PRIMARY OUTCOMES:
Mortality rate in the ketogenic group diet vs standard one | Up to nine months
Access in Intensive Care Unit in the ketogenic group diet vs standard one | Up to nine months
Need of Non Invasive Ventilation in the ketogenic group diet vs standard one | Up to nine months
Combined endpoint "mortality, ICU transfer or need for CPAP or intubation" in the ketogenic group diet vs standard one | Up to nine months

CONTACTS AND LOCATIONS:
Locations (1):
- Samir Giuseppe Sukkar, Genova, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mehta P, McAuley DF, Brown M, Sanchez E, Tattersall RS, Manson JJ; HLH Across Speciality Collaboration, UK. COVID-19: consider cytokine storm syndromes and immunosuppression. Lancet. 2020 Mar 28;395(10229):1033-1034. doi: 10.1016/S0140-6736(20)30628-0. Epub 2020 Mar 16. No abstract available. PMID 32192578
- [Background] Chen N, Zhou M, Dong X, Qu J, Gong F, Han Y, Qiu Y, Wang J, Liu Y, Wei Y, Xia J, Yu T, Zhang X, Zhang L. Epidemiological and clinical characteristics of 99 cases of 2019 novel coronavirus pneumonia in Wuhan, China: a descriptive study. Lancet. 2020 Feb 15;395(10223):507-513. doi: 10.1016/S0140-6736(20)30211-7. Epub 2020 Jan 30. PMID 32007143
- [Background] Karakike E, Giamarellos-Bourboulis EJ. Macrophage Activation-Like Syndrome: A Distinct Entity Leading to Early Death in Sepsis. Front Immunol. 2019 Jan 31;10:55. doi: 10.3389/fimmu.2019.00055. eCollection 2019. PMID 30766533
- [Background] Yoshikawa T, Hill T, Li K, Peters CJ, Tseng CT. Severe acute respiratory syndrome (SARS) coronavirus-induced lung epithelial cytokines exacerbate SARS pathogenesis by modulating intrinsic functions of monocyte-derived macrophages and dendritic cells. J Virol. 2009 Apr;83(7):3039-48. doi: 10.1128/JVI.01792-08. Epub 2008 Nov 12. PMID 19004938
- [Background] Ksiazek TG, Erdman D, Goldsmith CS, Zaki SR, Peret T, Emery S, Tong S, Urbani C, Comer JA, Lim W, Rollin PE, Dowell SF, Ling AE, Humphrey CD, Shieh WJ, Guarner J, Paddock CD, Rota P, Fields B, DeRisi J, Yang JY, Cox N, Hughes JM, LeDuc JW, Bellini WJ, Anderson LJ; SARS Working Group. A novel coronavirus associated with severe acute respiratory syndrome. N Engl J Med. 2003 May 15;348(20):1953-66. doi: 10.1056/NEJMoa030781. Epub 2003 Apr 10. PMID 12690092
- [Background] Kindler E, Thiel V. SARS-CoV and IFN: Too Little, Too Late. Cell Host Microbe. 2016 Feb 10;19(2):139-41. doi: 10.1016/j.chom.2016.01.012. PMID 26867172
- [Background] Channappanavar R, Fehr AR, Vijay R, Mack M, Zhao J, Meyerholz DK, Perlman S. Dysregulated Type I Interferon and Inflammatory Monocyte-Macrophage Responses Cause Lethal Pneumonia in SARS-CoV-Infected Mice. Cell Host Microbe. 2016 Feb 10;19(2):181-93. doi: 10.1016/j.chom.2016.01.007. PMID 26867177
- [Background] Huang C, Wang Y, Li X, Ren L, Zhao J, Hu Y, Zhang L, Fan G, Xu J, Gu X, Cheng Z, Yu T, Xia J, Wei Y, Wu W, Xie X, Yin W, Li H, Liu M, Xiao Y, Gao H, Guo L, Xie J, Wang G, Jiang R, Gao Z, Jin Q, Wang J, Cao B. Clinical features of patients infected with 2019 novel coronavirus in Wuhan, China. Lancet. 2020 Feb 15;395(10223):497-506. doi: 10.1016/S0140-6736(20)30183-5. Epub 2020 Jan 24. PMID 31986264
- [Background] Li B, Yang J, Zhao F, Zhi L, Wang X, Liu L, Bi Z, Zhao Y. Prevalence and impact of cardiovascular metabolic diseases on COVID-19 in China. Clin Res Cardiol. 2020 May;109(5):531-538. doi: 10.1007/s00392-020-01626-9. Epub 2020 Mar 11. PMID 32161990
- [Background] Ruan Q, Yang K, Wang W, Jiang L, Song J. Clinical predictors of mortality due to COVID-19 based on an analysis of data of 150 patients from Wuhan, China. Intensive Care Med. 2020 May;46(5):846-848. doi: 10.1007/s00134-020-05991-x. Epub 2020 Mar 3. No abstract available. PMID 32125452
- [Background] Tate RM, Repine JE. Neutrophils and the adult respiratory distress syndrome. Am Rev Respir Dis. 1983 Sep;128(3):552-9. doi: 10.1164/arrd.1983.128.3.552. No abstract available. PMID 6351681
- [Background] Keatings VM, Barnes PJ. Granulocyte activation markers in induced sputum: comparison between chronic obstructive pulmonary disease, asthma, and normal subjects. Am J Respir Crit Care Med. 1997 Feb;155(2):449-53. doi: 10.1164/ajrccm.155.2.9032177.
- [Background] Foucher P, Heeringa P, Petersen AH, Huitema MG, Brouwer E, Tervaert JW, Prop J, Camus P, Weening JJ, Kallenberg CG. Antimyeloperoxidase-associated lung disease. An experimental model. Am J Respir Crit Care Med. 1999 Sep;160(3):987-94. doi: 10.1164/ajrccm.160.3.9807139. PMID 10471629
- [Background] Johnson KJ, Fantone JC 3rd, Kaplan J, Ward PA. In vivo damage of rat lungs by oxygen metabolites. J Clin Invest. 1981 Apr;67(4):983-93. doi: 10.1172/jci110149. PMID 6894154
- [Background] Haegens A, Vernooy JH, Heeringa P, Mossman BT, Wouters EF. Myeloperoxidase modulates lung epithelial responses to pro-inflammatory agents. Eur Respir J. 2008 Feb;31(2):252-60. doi: 10.1183/09031936.00029307. Epub 2007 Dec 5. PMID 18057061
- [Background] van der Veen BS, de Winther MP, Heeringa P. Myeloperoxidase: molecular mechanisms of action and their relevance to human health and disease. Antioxid Redox Signal. 2009 Nov;11(11):2899-937. doi: 10.1089/ars.2009.2538. PMID 19622015
- [Background] Niu S, Bian Z, Tremblay A, Luo Y, Kidder K, Mansour A, Zen K, Liu Y. Broad Infiltration of Macrophages Leads to a Proinflammatory State in Streptozotocin-Induced Hyperglycemic Mice. J Immunol. 2016 Oct 15;197(8):3293-3301. doi: 10.4049/jimmunol.1502494. Epub 2016 Sep 12. PMID 27619992
- [Background] Van der Zwan LP, Scheffer PG, Dekker JM, Stehouwer CD, Heine RJ, Teerlink T. Hyperglycemia and oxidative stress strengthen the association between myeloperoxidase and blood pressure. Hypertension. 2010 Jun;55(6):1366-72. doi: 10.1161/HYPERTENSIONAHA.109.147231. Epub 2010 Apr 12. PMID 20385972
- [Background] Brennan ML, Penn MS, Van Lente F, Nambi V, Shishehbor MH, Aviles RJ, Goormastic M, Pepoy ML, McErlean ES, Topol EJ, Nissen SE, Hazen SL. Prognostic value of myeloperoxidase in patients with chest pain. N Engl J Med. 2003 Oct 23;349(17):1595-604. doi: 10.1056/NEJMoa035003. PMID 14573731
- [Background] Baldus S, Heeschen C, Meinertz T, Zeiher AM, Eiserich JP, Munzel T, Simoons ML, Hamm CW; CAPTURE Investigators. Myeloperoxidase serum levels predict risk in patients with acute coronary syndromes. Circulation. 2003 Sep 23;108(12):1440-5. doi: 10.1161/01.CIR.0000090690.67322.51. Epub 2003 Sep 2. PMID 12952835